CLINICAL TRIAL: NCT02648139
Title: A Randomized, Controlled, Double-blind Clinical Trial of a Eugenia Uniflora Linn. (Surinam Cherry) Dentifrice With Anti-gingivitis Properties
Brief Title: A Randomized, Controlled, Double-blind Clinical Trial of Surinam Cherry Dentifrice With Anti-gingivitis Properties
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Irlan de Almeida Freires, PhD, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Eugenia Dentifrice
Record Dates: First submitted 2016-01-05; First posted 2016-01-06 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis | interventions — Dentifrices

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental dentifrice (Experimental): Dentifrice containing the extract of Eugenia uniflora rip fruit. Each 10 ml of E. uniflora L. dentifrice comprises the following components: Hydroalcoholic extract of the ripe fruit of E. uniflora L. (3.0%), preservatives (parabens; 0.02 g), and dentifrice base (silicon dioxide, sodium lauryl sulfate, white dye, aromatic compounds, sodium saccharin, and Gangrez sodium salt; q.s.p.). Intervention protocol: three times per day (pea-like amount), for seven consecutive days.
  Interventions: Drug: Dentifrice
- Control Dentifrice (Active Comparator): Control dentifrice - Colgate total 12 (fluoride, 1500 ppm and triclosan, 0.3%)
  Intervention protocol: three times per day (pea-like amount), for seven consecutive days.
  Interventions: Drug: Dentifrice

INTERVENTIONS:
Drug: Dentifrice — 3x/day for 7 days.
  Other Names: Surrinam cherry dentifrice, Colgate total 12

SUMMARY:
In the present randomized, controlled, double-blind clinical trial, we investigated the short term clinical efficacy of a dentifrice containing Eugenia uniflora L. ripe fruit extract in preventing gingivitis in children.

DETAILED DESCRIPTION:
This was a randomized, controlled, double-blind clinical trial investigating the short term clinical efficacy of a dentifrice containing Eugenia uniflora L. ripe fruit extract in preventing gingivitis in children. The study consisted of a sample of 50 male and female subjects between the ages of 10 and 12 years old, who had clinical signs of gingivitis. The subjects were randomly assigned to one of two groups. The intervention group comprised 25 subjects who used the dentifrice with E. uniflora L. ripe fruit hydroalcoholic extract, three times per day, for seven consecutive days. The control group comprised 25 subjects who used the control dentifrice (fluoride, 1500 ppm and triclosan, 0.3%) for seven consecutive days.

The sample size was estimated using Fleming's single-stage procedure for phase II trials. With regard to the primary outcome, a response proportion of at least 50% was defined as being clinically significant. The type I error was set as 0.05, and the type II error was set at 0.1. Based on these values, a sample size of 20 individuals per trial arm would provide 90% power (1-β) to detect any clinically relevant treatment difference of 50% or greater compared to baseline. Taking into consideration an attrition rate of approximately 20%, the final sample size per trial arm comprised 25 individuals.

Clinical examinations were performed at baseline and after seven days of dentifrice use. The examination was performed by a single examiner who was adequately calibrated with a Kappa statistic of 0.8, which is considered to be satisfactory agreement according to Landis & Koch. The examination data were recorded in a specific clinical chart. The diagnosis of gingivitis (primary outcome) was assessed using the Gingival Bleeding Index (GBI) proposed by Ainamo and Bay. The accumulation of biofilm (secondary outcome) was assessed with the Simplified Oral Hygiene Index (OHI-S) described by Greene and Vermilion. Prior to the study, all of the subjects were instructed on correct tooth brushing techniques and received a kit that contained a toothbrush and one of the dentifrices (without the identification of its contents). The dentifrices were also masked with regard to flavor and color so that they could not be identified. In addition, the examiner had no knowledge of the subject allocation. Thus, the study was double-blind.

The sample included only subjects who had not used an antimicrobial in the last two months, including topical fluoride.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 10 to 12 years old with clinical signs of gingivitis (bleeding on probing);
* Presence of at least 20 dental elements
* Not using orthodontic fixed appliances
* Susceptibility to form biofilm and gingival inflammation
* Absence of systemic disease

Exclusion Criteria:

- Subjects who had used an antimicrobial in the last two months, including topical fluoride.

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2008-12; Primary Completion 2010-02 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Reduction in gingivitis levels | Baseline and seven days
  The primary outcome of interest was the reduction in the levels of gingivitis (bleeding on probing) assessed by the Gingival Bleeding Index (GBI) proposed by Ainamo and Bay.

SECONDARY OUTCOMES:
Reduction in the amount of plaque | Baseline and seven days
  The secondary outcome of interest was the reduction in the amount of plaque assessed by the Simplified Oral Hygiene Index (OHI-S) described by Greene and Vermilion.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo D Castro, PhD, Principal Investigator — Federal University of Paraíba